CLINICAL TRIAL: NCT04549974
Title: Characterization of the Increase and Distribution of Myocardial Blood Flow During Heat Exposure
Brief Title: Characterization of Myocardial Blood Flow During Heat Exposure
Acronym: PET-Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Daniel Gagnon, Principal Investigator, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICM 2020-2719
Record Dates: First submitted 2020-08-25; First posted 2020-09-16 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Hot Weather; Adverse Effect; Healthy; Coronary Artery Disease; Aging
Keywords: Heat; PET imaging; Myocardial blood flow
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive heat exposure (Experimental)
  Interventions: Other: Heat exposure

INTERVENTIONS:
Other: Heat exposure — Participants will be exposed to heat exposure via a water-perfused suit to increase internal body temperature by 1.5 degrees Celsius.

SUMMARY:
The purpose of this study is to determine the increase in myocardial blood flow during heat exposure and how this response is affected by age and coronary artery disease.

DETAILED DESCRIPTION:
As a result of climate change, heat waves are more frequent and of longer duration. These heat waves are associated with a higher risk of hospitalization and mortality in vulnerable populations such as people with cardiovascular disease or cardiovascular risk factors. It has been hypothesized that this observation may be explained by the cardiovascular demands imposed by heat exposure.

Heat exposure requires increased cardiac work that may place individuals with cardiovascular disease at risk of ischemic events if the metabolic demand is not compensated by adequate blood supply. However, the extent to which cardiac work increases during heat exposure remains unknown. The aim of this study is to test the hypothesis that heat exposure increases myocardial blood flow and that this increase is affected by age and coronary artery disease.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* Age between 18-40 years or 60-80 years
* Non-smoker (≥1 year)
* Non-diabetic
* Normal kidney function
* Body Mass Index <30 kg/m2
* Resting blood pressure <140/<90 mmHg
* Resting heart rate <100 bpm

Inclusion Criteria for Participants with Coronary Artery Disease:

* Age between 60-80 years old
* History of angiographic coronary disease (≥70% arterial diameter narrowing of at least one major epicardial coronary artery) and/or prior coronary revascularization and/or documented prior acute coronary syndrome and/or perfusion defect during stress testing
* Stable medications (≥4 weeks) prior to enrollment

Exclusion Criteria for Healthy Participants:

* Diagnosis of heart, vascular, respiratory, neurological or metabolic disease and/or a prescription of medication for the treatment of these diseases
* Pregnancy or lactation
* Dyslipidemia not controlled by medication

Exclusion Criteria for Participants with Coronary Artery Disease:

* Recent hospitalization (<3 months) related to coronary artery disease
* Unstable angina (<3 months)
* Recent coronary artery bypass surgery (<3 months)
* Left branch block
* Ejection fraction <40% and/or clinical signs of heart failure
* Severe valvular heart disease
* Hypertension not controlled by medication
* Diabetes not controlled by medication and/or serious complications related to diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Global myocardial blood flow | Change from baseline to an increase in internal body temperature of 1.5 degrees Celsius, estimated average = 90 minutes
  Measured by PET imaging with 82rubidium

SECONDARY OUTCOMES:
Myocardial blood flow distribution | Change from baseline to an increase in internal body temperature of 1.5 degrees Celsius, estimated average = 90 minutes
  Measured by PET imaging with 82rubidium
Heart rate | Change from baseline to an increase in internal body temperature of 1.5 degrees Celsius, estimated average = 90 minutes
  Measured by electrocardiogram
Systolic and diastolic blood pressure | Change from baseline to an increase in internal body temperature of 1.5 degrees Celsius, estimated average = 90 minutes
  Measured by automated auscultation of the brachial artery
Body weight | Measured before and after heat exposure, estimated average = 120 minutes
  Measured with a scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gagnon, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barry H, Iglesies-Grau J, Chaseling GK, Paul J, Gosselin C, D'Oliviera-Sousa C, Juneau M, Harel F, Kaiser D, Pelletier-Galarneau M, Gagnon D. The Effect of Heat Exposure on Myocardial Blood Flow and Cardiovascular Function. Ann Intern Med. 2024 Jul;177(7):901-910. doi: 10.7326/M24-3504. Epub 2024 Jun 11. PMID 38857500